CLINICAL TRIAL: NCT04476940
Title: An Intervention to Promote COVID-19 Breastfeeding Guideline Adherence Among African American Mothers
Brief Title: COVID-19 Breastfeeding Guideline for African-Americans
Acronym: COVID-BF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Meharry Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 330875
Record Dates: First submitted 2020-07-13; First posted 2020-07-20 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Covid19; Exclusive Breastfeeding
Keywords: COVID-19; Exclusive Breastfeeding; Breastfeeding Guidelines; African American
MeSH Terms: conditions — COVID-19; Breast Feeding

STUDY DESIGN:
Intervention Model Description: Pre-Test Post-test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COVID BF-Support (Experimental): COVID-19 breastfeeding guideline education and support for pregnant women.
  Interventions: Behavioral: COVID-19 Breastfeeding Support

INTERVENTIONS:
Behavioral: COVID-19 Breastfeeding Support — Intervention will be implemented by trained prenatal care providers to provide comprehensive exclusive breastfeeding and COVID-19 breastfeeding guideline education and support to study participants.

SUMMARY:
Newborns and infants receive passive natural immunity through maternal antibodies present in breastmilk to fight infections caused by viruses such as the COVID-19, until they develop active immunity by illness or vaccination. Such immunity will become the main stay for preventing future waves of COVID-19 epidemics. The high COVID-19 mortality among African Americans is ascribed partly to compromised immune status associated with comorbidity. Exclusive breastfeeding (EBF) is the effective low-cost natural strategy for building immunity right from birth. African Americans record the lowest EBF rates and also lack workplace support. This intervention includes a 10-hour course extracted from 90-hour CLC online program, sufficient to prepare physicians to partner with certified lactation consultant (CLC) to provide their patients comprehensive COVID-19 breastfeeding guidelines, training, and support to afford their babies the benefits of breastmilk antibodies, the best line of defense against COVID-19, until availability of safe vaccines. The Breastfeeding Report Card indicates slow improvements in overall breastfeeding rates with persisting disparities. Improving EBF rates can contribute to increased COVID-19 immunity among infants. Preliminary data in Nashville indicates excellent breastfeeding benefit knowledge and intent, but limited training to succeed. Hospital staff encourage breastfeeding but routinely offer formula at birth. Most physicians who provide prenatal care do not actively promote breastfeeding nor routinely offer CLC referral. This single action by physicians can halt routines that compromise successful EBF. The program long-term goal is to prepare obstetricians to actively promote comprehensive breastfeeding among African American mothers. The immediate objective is to develop and evaluate feasibility and effectiveness of an intervention designed to increase COVID-19 breastfeeding guideline adherence and improve EBF skills and rates among African American mothers. The rationale is that mothers who receive physician prenatal encouragement and CLC referral will make confident informed decisions, adopt COVID-19 breastfeeding guidelines, safely meet their EBF goals, and provide their infants with appropriate antibodies. The expected outcome is that patient participants will adhere to COVID-19 breastfeeding guidelines and record 3-month EBF rate 60 percent or greater.

DETAILED DESCRIPTION:
Phase 1: COVID-19 Breastfeeding Guideline Assessment Survey. 40 mothers who delivered during the period starting from January 1, 2020 to date will be recruited and consented to assess their exclusive breastfeeding (EBF) and COVID-19 breastfeeding patterns using a survey designed to be completed by interview on Zoom, phone, or any other social-distancing platform. Information to be collected in this survey will include: demography, medical history, COVID-19 status; COVID-19 breastfeeding guideline action; Stay-home pattern; Breastfeeding frequency and duration; Breastmilk expression frequency/duration; Frequency and volume of feeds with expressed breastmilk or formula.

Phase 2: Intervention Development:

Participating physicians will attend two 2-hour Zoom sessions, a 4-Module Online Breastfeeding Course, and a 1-hour orientation Zoom session in groups of not more than ten. The following presentations, course, surveys, other materials to be developed:

1. . Three presentations: i). Introduction: Healthy People 2020 Breastfeeding Objectives, Tennessee breastfeeding statistics, Breastfeeding role of physicians, nurses, and certified lactation consultants (CLC). ii). Breastfeeding Challenges Faced by Mothers. iii). Obstetrician Breastfeeding Promotion Challenges.
2. . Online Breastfeeding Promotion 101: A 10-hour course to be developed in partnership with Breastfeeding OUTLOOK, an online continuing education provider.
3. . Research Tools: COVID-19 Breastfeeding Guideline Assessment surveys; Pre- and Post-Intervention surveys for physicians; Pre- and Post-Intervention surveys for patients; Consent forms for physicians; Consent and HIPAA forms for patients; Recruitment flyer and Breastfeeding brochure for patients.
4. . Moderator Script for Community Engagement to guide the community-patient-provider stakeholder community advisory board (CAB) discussion sessions to review and make recommendations for revision to the following: intervention program, consent forms, surveys, brochure, COVID-19 related guidelines for pregnant and lactating mothers, and strategies to enhance participation. The 12-Person CAB of 4 mothers, 2 nurses/midwives, 2 CLCs, 2 physicians, a virologist, and a community leader. Investigator obstetrician Ladson, G. will be the moderator and the CAB recorder will be investigator Britt, A.

Phase 3: Program Implementation Feasibility and Evaluation:

20 Obstetricians/Physicians will be consented and enrolled to participate as program providers, and expected to complete the following 5 tasks:

1. . Pre-Intervention Survey: This is 15-minute self-administered pre-test survey to capture breastfeeding promotion knowledge and practices, and COVID-19, other disease, and drug related breastfeeding guidelines.
2. . First In-Person Session: 2-hour Zoom session in groups of not more than 10 participants to disseminate Program introduction (20 minutes); Breastfeeding challenges faced by mothers (40 minutes); Obstetrician breastfeeding promotion challenges (40 minutes); Closing session (20 minutes) for Concerns, Q & A.
3. . Online Breastfeeding Course 101: Participant physicians will enroll in Breastfeeding OUTLOOK and complete a 10-hour module over a two-week period.
4. . Second In-Person Session: 2-hour Zoom session in groups of 10 to provide intervention guidelines, research strategies and skills for participant recruitment, consenting, and survey administration by interview.
5. . Intervention Implementation: 20 physicians will each be expected to recruit 10 study participants in the third trimester of pregnancy from their prenatal clients over a period of two months. Physicians will complete a pre-intervention survey at enrollment and post-intervention survey 8 months after enrollment in the program. The physicians will receive intervention protocol, patient HIPPA & consent forms, flyers, and survey booklet after signed consent received by email, and attend a one-hour program orientation in company of an office staff and/or resident physician scheduled in groups of four. The 200 study participants will sign informed consent, complete a pre-intervention patient survey, continue prenatal care, and will be followed up at 1-month and at 3-months postpartum to complete the post-intervention patient survey.

Study Questionnaires. i) Mother COVID-19 Breastfeeding Guideline Assessment Survey: Demography, medical history, items from Centers for Disease Prevention and Control (CDC) & Baby-Friendly Hospital Initiative (BFHI) breastfeeding surveys, EBF pattern since January 1, 2020, COVID-19 guideline items, COVID-19 status, Stay-home history.

ii) Physician pre-intervention survey: Monthly prenatal volume, breastfeeding knowledge, and practices, CLC referral pattern, COVID-19 and other disease specific EBF guidelines.

iii) Physician post-intervention survey: Breastfeeding knowledge and practices, COVID-19 and other disease specific EBF guidelines. Number of participants enrolled and number of CLC referrals.

iv) Patient pre-intervention survey: Demography, medical history, CDC & BFHI breastfeeding survey items, physician interaction items, previous CLC encounter, COVID-19 guideline items, COVID-19 status, Stay-home history.

v) Patient post-intervention survey: CLC referral, CLC appointment and breastfeeding class attendance; COVID-19 guideline adherence; EBF initiation, frequency/duration of EBF; frequency and duration of breastmilk expression (manual or pump); frequency and volume of formula or breastmilk feeds. Infant feeding and growth pattern from medical records and growth charts. COVID-19 serology test (optional).

ELIGIBILITY:
Inclusion Criteria:

* Assessment Survey: Mothers who had a baby in 2020.
* Intervention Participants: Women in late 2nd or 3rd pregnancy trimester enrolled for prenatal care by participating physicians.

Exclusion Criteria:

* Assessment Survey: Mothers who had a baby prior to 2020.
* Intervention Participants: Not pregnant, in 1st trimester of pregnancy, not enrolled for prenatal care by participating physician.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
COVID-19 breastfeeding guidance adherence at birth. | At birth.
  Percentage of participants who recorded an adherence score of 4 and above during the first week of birth.
  Range: 0 to 100.
COVID-19 breastfeeding guidance adherence at 1-month postpartum. | At 1-month postpartum.
  Percentage of participants who recorded an adherence score of 4 and above at 1-month postpartum.
  Range: 0 to 100.
COVID-19 breastfeeding guidance adherence at 3-months postpartum. | At 3-months postpartum.
  Percentage of participants who recorded an adherence score of 4 and above at 3-months postpartum.
  Range: 0 to 100.
Exclusive breastfeeding at birth. | At birth.
  Percentage of participants who exclusively breastfed at birth. Range: 0 - 100.
Exclusive breastfeeding at 1-month. | At 1-month.
  Percentage of participants who exclusively breastfed at 1-month postpartum. Range: 0 - 100.
Exclusive breastfeeding at 3-months. | At 3-months.
  Percentage of participants who exclusively breastfed at 3-months postpartum. Range: 0 - 100.

SECONDARY OUTCOMES:
COVID_Status | 3-months postpartum
  Infant COVID-19 test: Positive or Negative
COVID-19 Immunoglobulin G | 3-months postpartum
  Infant COVID-19 Immunoglobulin G serology test result.
COVID-19 Immunoglobulin M | 3-months postpartum
  Infant COVID-19 Immunoglobulin M serology test result.

OTHER OUTCOMES:
Certified Lactation Consult in pregnancy. | At Birth.
  Percentage of patients who consulted a Certified Lactation Consultant before delivery.
  Range: 0 - 100
Certified Lactation Consult after delivery. | At 1-month postpartum.
  Percentage of patients who consulted a Certified Lactation Consultant up to 1-month postpartum.
  Range: 0 - 100
COVID-19 breastfeeding guideline knowledge score change. | 1-month postpartum
  Change in pre- and post-intervention COVID-19 breastfeeding guideline knowledge score stratified to "Low" & "High".

CONTACTS AND LOCATIONS:
Overall Officials: Samuel E Adunyah, Ph.D., Study Director — Meharry Medical College; Carlton Z Adams, M.D., Study Chair — Meharry Medical College; Flora A Ukoli, M.D., MPH., Principal Investigator — Meharry Medical College
Locations (1):
- Meharry Medical College, Nashville, Tennessee, United States